CLINICAL TRIAL: NCT07274345
Title: Prevalence and Risk Factors Associated With Resistance to Antiviral Therapy in Egyptian Patients With Chronic Hepatitis B Virus Infection
Brief Title: Prevalence and Risk Factors of Antiviral Resistance in Egyptian HBV Patients
Acronym: PRARE-CHB
Status: Not yet recruiting | Type: Observational
Sponsor: Amira Mohamed Zidan (Other)
Responsible Party: Sponsor-Investigator, Amira Mohamed Zidan, Resident Doctor Tropical Medicine and Gastroenterology, Sohag University
Organization: Sohag University (Other)
Other Study IDs: Soh-Med--25-11-5MS
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Chronic Hepatitis B - Antiviral Drug Resistance - Hepatitis B Virus (HBV) Infection
MeSH Terms: conditions — Hepatitis B; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- This cohort includes adult Egyptian patients diagnosed with chronic hepatitis B virus (HBV) infectio

SUMMARY:
This study aims to determine the prevalence of antiviral drug resistance among Egyptian patients with chronic hepatitis B virus (HBV) infection and to identify the associated demographic, clinical, and virological risk factors. Understanding patterns of resistance will help improve treatment selection and optimize long-term management strategies for HBV patients.

ELIGIBILITY:
Inclusion Criteria:

* This study will include all chronic HBV-infected patients, either cirrhotic or not, receiving TDF 300 mg, ETV 0.5 or 1mg, or lamivudine 100 mg, irrespective of HBeAg status. The HBV chronicity is defined by persistence of HbsAg positivity for more than 6 months.

Exclusion Criteria:

* Patients younger than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Egyptian patients diagnosed with chronic hepatitis B virus (HBV) infection and receiving antiviral therapy in routine clinical practice. Participants are recruited from outpatient hepatology and gastroenterology clinics and represent a real-life population of treated chronic HBV patients.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients Exhibiting Antiviral Resistance Detection of HBV Antiviral Resistance Mutations | 6 months

IPD SHARING:
Plan to Share IPD: Undecided